CLINICAL TRIAL: NCT04001400
Title: Treatment Response of High-dose and Standard-dose Rabeprazole for Gastroesophageal Reflux Disease With Extra-esophageal Manifestations: a Single-center, Randomized, Open-label Trial.
Brief Title: Treatment Response of High-dose and Standard-dose Rabeprazole for Extra-esophageal Reflux.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Principal Investigator, Dong Ho Lee, Director, Clinical Research, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-DHLIDRA
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Esophageal Disease
Keywords: Gastroesophageal Reflux
MeSH Terms: conditions — Esophageal Diseases; Gastroesophageal Reflux | interventions — Rabeprazole; BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose rabeprazole (Experimental): Rabeprazole 20mg twice daily by mouth before breakfast and dinner for 8 weeks
  Interventions: Drug: Rabeprazole 20mg bid
- Standard-dose rabeprazole (Active Comparator): Rabeprazole 20mg once daily by mouth before breakfast for 8 weeks
  Interventions: Drug: Rabeprazole 20mg qd

INTERVENTIONS:
Drug: Rabeprazole 20mg bid — Rabeprazole 20mg tablet b.i.d.
  Other Names: Rabiet
  Arms: High-dose rabeprazole
Drug: Rabeprazole 20mg qd — Rabeprazole 20mg tablet q.d.
  Other Names: Rabiet
  Arms: Standard-dose rabeprazole

SUMMARY:
This is a single-center, randomized, open-label clinical study to assess the treatment response of high-dose rabeprazole compared with standard-dose rabeprazole in patients with extra-esophageal manifestations of gastroesophageal reflux disease.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease is a condition in which reflux of stomach contents into the esophagus. This disease can be classified in to two subtypes according to the symptoms; Typical symptoms such as heartburn and regurgitation, and atypical symptoms (extra-esophageal symptoms) such as chronic cough, asthma, non-cardiac chest pain, globus sensation, etc.

Acid suppression with proton pump inhibitors is the mainstream of therapy for the extra-esophageal manifestation as well as the typical symptoms of gastroesophageal reflux disease.

However, there is controversy about the efficacy of proton pump inhibitors on extra-esophageal reflux.

Therefore, we aimed to assess the effect of proton pump inhibotor (rabeprazole) on the extra-esophageal manifestation of gastroesophageal reflux disease, through comparison of treatment response with high-dose and standard-dose rabeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Age is over 20 years old, under 80 years old, men or women
* Patients who had experienced extra-esophageal symptoms of gastroesophageal reflux disease more than once a week within the last month prior to the start of the study

Exclusion Criteria:

* Patients administered with prokinetics, H2 receptor antagonists, proton pump inhibitors, anticholinergic drugs or non-steroid anti-inflammatory drugs prior to study in 4 weeks
* Patients administered with anti-thrombotic drugs
* Patients taking other investigational drugs or participating in other clinical studies in 4 weeks
* Patients with esophageal stricture, esophageal varix, Barrett's esophagus, peptic ulcer or gastrointestinal bleeding
* Patients with Zollinger-Ellison syndrome
* Patients with any kind of malignant tumor
* Patients with surgery related to gastroesophageal
* Patients with significant cardiovascular, pulmonary, heptic, renal, hemopoietic or endocrine system primary disease
* Patients with neuropsychiatric disorder, alcoholism, or drug abuse
* Women either pregnant or breast feeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2014-05-21 (Actual); Study Completion 2014-05-21 (Actual)

PRIMARY OUTCOMES:
Effective improvement of symptoms | 8 weeks
  A percentage of subjects showed effective improvement of extra-esophageal symptoms of gastroesophageal reflux disease by assessing the average sum of the questionnaire symptom scores.
  The definition of "effective improvement" is the subjects showed ≥50% reduction from the initial questionnaire score.
  The symptom questionnaire consists of a 5-graded Likert scale for each symptom to assess intensity of symptoms.
  [score 0: no symptoms, score 1: mild symptoms that is not easily felt, score 2: moderate symptoms but not affect daily life, score 3: severe symptoms that hinder daily life or sleep, score 4: very severe symptoms that cannot lead to normal daily life or sleep]
  In this trial, extra-esophageal symptoms consist of eight symptoms; non-cardiac chest pain, cough, globus, wheezing, laryngopharyngitis, hoarseness, belching and dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ho Lee, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bungdang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho JH, Shin CM, Yoon H, Park YS, Kim N, Lee DH. Efficacy of a high-dose proton pump inhibitor in patients with gastroesophageal reflux disease: a single center, randomized, open-label trial. BMC Gastroenterol. 2020 Aug 18;20(1):275. doi: 10.1186/s12876-020-01410-z. PMID 32811427